CLINICAL TRIAL: NCT02298569
Title: Early Postnatal Discharge in a French Perinatal Network
Acronym: SORPRISE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Réseau Périnatal Alpes-Isere (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DCIC 13 17
Record Dates: First submitted 2014-08-29; First posted 2014-11-24 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Pregnancy Complications Nos; Labor/Delivery Problems Nos; Vitality; Newborn
Keywords: patient discharge; hospital readmission; postnatal care; Home Care Services; Cost-Benefit Analysis; Personal satisfaction; Community Care Networks
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase 1 (before multi-pronged program) (No Intervention): 400 low-risk mothers having given birth without any complication to a healthy newborn are to be recruited in the 5 maternity wards of a French perinatal network consecutively, whatever the duration of their hospital stay
- Phase 2 (after multi-pronged program) (Experimental): 400 low-risk mothers having given birth without any complication to a healthy newborn are to be recruited in the 5 maternity wards of the same French perinatal network 3 months after the intervention (introduction of the multi-pronged program) consecutively, whatever the duration of their hospital stay
  Interventions: Behavioral: multi-pronged program to improve early postpartum discharge

INTERVENTIONS:
Behavioral: multi-pronged program to improve early postpartum discharge — Better team integration and changes to promote interprofessional collaboration and communication between healthcare providers involved in pre- and post-natal care in a perinatal network.
  Transition optimization: all involved healthcare professionals will complete a specific form during pregnancy and hospitalization to coordinate support safe process, and to improve quality transitions to outpatient midwives and pediatrician. A check-list will be completed by the mother to assess whether she agrees to early discharge and that she is aware of its conditions Implementation of best practices about early discharge after delivery to improve safety of early discharge particularly for neonates at risk (jaundice and dehydration).
  Other Names: team integration and culture change; transition optimisations; implementation of best practices
  Arms: Phase 2 (after multi-pronged program)

SUMMARY:
The purpose of this "before-after" study is to determine the effectiveness of a multidimensional intervention to increase the rate for early discharge of low-risk mothers and the healthy newborn in a perinatal network.

DETAILED DESCRIPTION:
In March 2014, the French Health Authorities edited new guidelines about early discharge after delivery. Early discharge is defined as a discharge during the 72 hours following vaginal delivery of low-risk mothers and their healthy newborn. These guidelines defined the conditions of eligibility for early discharge for mothers and babies, and the different criteria of their follow-up at home by midwives .

The average length of stay following normal delivery is higher in France than in other European countries: eg : 4.3 days in France vs 2.2 days in Sweden (OECD indicators 2011) On the other hand, according to an investigation conducted by a patients association, 38% women declared that they felt that their hospitalization was too long after their baby's birth, but their request for a shorter stay had not been taken into account by hospital caregivers. The investigators hypothesis is that the rate of early discharge could be increased by a multi-pronged program coordinated in a perinatal network, and could improve quality of postpartum care, and women's satisfaction.

The "Réseau Périnatal Alpes Isère" is a perinatal network located in French Alps region. Its purpose is to coordinate 5 maternity services an organization of midwives providing pre and postnatal home care, for about 10000 births annually. In 2010, according to the hospital database provided by the Medical Information Systems Program, early discharge concerned only 4.1% of mothers between 0 and 48 hours after delivery . At the same time, 65% of women could be considered as at low risk, considering they gave birth to a healthy singleton, born after 38 weeks of gestation by vaginal delivery. This rate is not precise, in view of the lack of availability of documented rate of non-eligibility for early discharge such as non- eutrophic babies, or adverse events during postpartum and the neonatal period.

ELIGIBILITY:
Inclusion Criteria:

"1" low risk mothers ith uncomplicated pregnancy and birth defined as

* lack of mental disability
* lack of referred problems about mother to infant bonding
* lack of precarious state
* vaginal delivery without bleeding more than 500cc
* lack of postpartum complications during hospitalization

"2" low risk baby defined as

* singleton
* gestational age >= 38 weeks
* apgar score > 7 at 5 minutes life
* normal weight expected for gestational age
* lack of infection, or jaundice

Exclusion Criteria:

* person deprived of liberty
* person who does not speak French
* person not covered by health insurance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-01 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
rate of early discharge | 15 days after delivery
  number of early postnatal discharges (2-72 hours after delivery) among eligible population: i.e. low risk mothers and low risk newborns, before and after a major change in the organization of integrated managed care, in a perinatal network. The rate of emergency medical consultations and or re-hospitalization for mothers and babies will be recorded among women who had an early postnatal discharge compared to women with standard hospital stay. Every eligible women will have a phone interview 15 days after delivery to assess the duration of hospitalization in the maternity ward and to report any emergency medical consultation or rehospitalization after discharge of mother and baby.

SECONDARY OUTCOMES:
rehospitalization or emergency visits for mothers and babies | from postnatal discharge up to 15 days after delivery
  number of rehospitalization or emergency medical visits for mothers and/or babies observed during the first 15 days after delivery, among the eligible population i.e. low risk mothers and low risk newborns, whatever the duration of their hospital stay. Every eligible women will have a phone interview 15 days after delivery to assess type of hospital discharge (early or standard), and if necessary, report any emergency medical consultation or rehospitalization after hospital discharge for baby and/or mother
continuation of breastfeeding | 60 days after delivery
  number of women continuing breastfeeding beyond 60 days postpartum, before and after intervention. Every women who had early postnatal discharge will have a phone interview 60 days after delivery to assess the duration of breastfeeding
maternal satisfaction | 45 days after delivery
  maternal satisfaction based on adapted WOMen's views of Birth Postnatal Satisfaction Questionnaire mean scores (WOMBSQ questionnaire). The WOMen's views of Birth Postnatal Satisfaction Questionnaire (WOMBSQ questionnaire) asks about quality of postnatal care provided both in the maternity ward during the hospital stay, and at home by the midwife during 2-4 days follow-up. The scores will be compared before and after the intervention. Every women who had early postnatal discharge, will be asked to complete the WOMen's views of Birth Postnatal Satisfaction Questionnaire form (on line or by post) 45 days after delivery
maternal depression | 45 days after delivery
  postnatal depression defined as a score higher than 12 on Edinburgh Postpartum Scale (EDPS) among women with early discharge from hospital will be compared before and after the intervention. Every women who had early postnatal discharge, will be asked to complete the EDPS form (on line or by post) 45 days after delivery to assess maternal depressive symptoms
maternal quality of life | 45 days after delivery
  mean scores of Short-Form Health Survey (SF-12) among women with early discharge from hospital to be compared before and after intervention. Every women who proceeded to early postnatal discharge, will be asked to complete SF-12 form (on line or by post) 45 days after delivery to asses maternal quality of life
satisfaction about the medical feed back after discharge | 45 - 60 days after delivery
  mean scores of satisfaction adapted from the questionnaire Satisfaction of the Patients at the Hospital in Region Aquitaine-Committee of evaluation 2009(SAPHORA-Committee of evaluation 2009) French form, about the quality of medical feedback after early discharge from hospital to be compared before and after intervention. Every community practitioner (general practitioner, paediatrician, midwife) who saw the mothers and baby during follow-up will be asked to complete a form , 45 or 60days after delivery to assess the quality of medical information given by the hospital to community practitioners, and the quality of the discharge summary
cost effectiveness | 15 days
  cost of early discharge, that is cost of hospitalization and cost of follow-up and cost of readmission to be compared with cost of routine hospitalization and eventual readmission for healthy mothers and babies, assessed during phone interviews with mothers
associated factors to early discharge | 15 days
  information about early discharge during pregnancy, socioeconomic factors, medical antecedents, type of prenatal follow-up, assessed by phone call interview with every eligible mother
compliance to french guidelines | 15 days
  compliance to French guidelines edited in 2014 about the organization of early discharge and home follow-up to be assessed by phone interview with midwife who performed home follow-up of mothers after early discharge
mother-infant bonding | 15 days after delivery
  mean Mother to Infant bonding scale (MIB score ) at 15 days after delivery, among eligible population that is low risk mothers and low risk newborns, whatever the duration of hospital stay. Every eligible women will get a form (on line or by post) 15 days after delivery to assess the feelings of mother towards their new baby. Mothers will be asked during the phone interview how they would like to complete this form : paper sent by post, or on line.

CONTACTS AND LOCATIONS:
Overall Officials: Claudine MARTIN, Principal Investigator — RPAI (Réseau Périnatal Alpes Isere), CHU Grenoble
Locations (5):
- France (5):
  - Clinique des Cèdres, Échirolles
  - Clinique Mutualiste, Grenoble
  - Hopital Couple Enfant, La Tronche
  - Clinique Belledonne, Saint-Martin-d'Hères
  - CH Voiron, Voiron

REFERENCES:
- [Background] Liu S. Rate of neonatal hospital readmission after discharge following birth. Canadian Perinatal Health Report 2003; 104-106. http://www.hc-sc.gc.ca/pphb-dgspsp/rhs-ssg/index.html
- [Background] Ellberg L, Hogberg U, Lundman B, Kallen K, Hakansson S, Lindh V. Maternity care options influence readmission of newborns. Acta Paediatr. 2008 May;97(5):579-83. doi: 10.1111/j.1651-2227.2008.00714.x. PMID 18394103
- [Background] Radmacher P, Massey C, Adamkin D. Hidden morbidity with "successful"early discharge.J Perinatol.2002;22:15-20 VIBoulvain M, Perneger TV, Othenin-Girard V, PetrouS, Berner M, Irion O. Home-based versus hospital-based postnatal care:arandomisedtrial.BJOG: an International Journal of Obstetrics and Gynaecology 2004; 111: 807-813.
- [Background] Oddie SJ, Hammal D, Richmond S, Parker L. Early discharge and readmission to hospital in the first month of life in the Northern Region of the UK during 1998: a case cohort study. Arch Dis Child. 2005 Feb;90(2):119-24. doi: 10.1136/adc.2003.040766. PMID 15665161
- [Background] Sainz Bueno JA, Romano MR, Teruel RG, Benjumea AG, Palacin AF, Gonzalez CA, Manzano MC. Early discharge from obstetrics-pediatrics at the Hospital de Valme, with domiciliary follow-up. Am J Obstet Gynecol. 2005 Sep;193(3 Pt 1):714-26. doi: 10.1016/j.ajog.2005.01.015. PMID 16150265
- [Background] Johansson K, Aarts C, Darj E. First-time parents' experiences of home-based postnatal care in Sweden. Ups J Med Sci. 2010 May;115(2):131-7. doi: 10.3109/03009730903431809. PMID 20074000
- [Background] Shaw E, Levitt C, Wong S, Kaczorowski J; McMaster University Postpartum Research Group. Systematic review of the literature on postpartum care: effectiveness of postpartum support to improve maternal parenting, mental health, quality of life, and physical health. Birth. 2006 Sep;33(3):210-20. doi: 10.1111/j.1523-536X.2006.00106.x. PMID 16948721
- [Background] Bravo P, Uribe C, Contreras A. Early postnatal hospital discharge: the consequences of reducing length of stay for women and newborns. Rev Esc Enferm USP. 2011 Jun;45(3):758-63. doi: 10.1590/s0080-62342011000300030. PMID 21710086
- [Background] http://www.sante.gouv.fr/IMG/pdf/Les_naissances_en_2010_et_leur_evolution_depuis_2003.pdf
- [Background] OCDE (2009), Panorama de la santé 2009 : Les indicateurs de l'OCDE, Éditions OCDE.doi : 10.1787/health_glance-2009-fr
- [Background] Smith LF. Postnatal care: development of a psychometric multidimensional satisfaction questionnaire (the WOMBPNSQ) to assess women's views. Br J Gen Pract. 2011 Oct;61(591):e628-37. doi: 10.3399/bjgp11X601334. PMID 22152835
- [Background] Antoniotti S, Baumstarck-Barrau K, Simeoni MC, Sapin C, Labarere J, Gerbaud L, Boyer L, Colin C, Francois P, Auquier P. Validation of a French hospitalized patients' satisfaction questionnaire: the QSH-45. Int J Qual Health Care. 2009 Aug;21(4):243-52. doi: 10.1093/intqhc/mzp021. Epub 2009 Jun 23. PMID 19549673
- [Background] Gandek B, Ware JE, Aaronson NK, Apolone G, Bjorner JB, Brazier JE, Bullinger M, Kaasa S, Leplege A, Prieto L, Sullivan M. Cross-validation of item selection and scoring for the SF-12 Health Survey in nine countries: results from the IQOLA Project. International Quality of Life Assessment. J Clin Epidemiol. 1998 Nov;51(11):1171-8. doi: 10.1016/s0895-4356(98)00109-7. PMID 9817135
- [Background] Edinburgh Depression Scale Translated Government of Western Australia Department of Health www.folkhalsoguiden.se/upload/Psykisk Hälsa/Edinburgh Depression Scale Translated Government of Western Australia Department of Health.pdf
- [Background] DOMECQ, S. AUSTRUY, J.VIOT, F. CADIOT, C POURIN. Evaluation de la satisfaction des correspondants externes : Rapport régional, mars 2009. CCECQA -Hôpital Xavier Arnozan -33604 Pessac www.ccecqa.asso.fr